CLINICAL TRIAL: NCT03996070
Title: Randomised, Sham Controlled Trial of Fotona Smooth Erbium Yag Laser In the Treatment of Stress Urinary Incontinence
Brief Title: VESPER: Stress Urinary Incontinence STUDY
Acronym: VESPER-SUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-FAM-01
Record Dates: First submitted 2019-03-28; First posted 2019-06-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Female Stress Incontinence
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Active Comparator): Therapeutic dose regime
  Interventions: Procedure: Laser therapy
- Sham arm (Placebo Comparator): Sub-therapeutic dose regime
  Interventions: Procedure: Laser therapy

INTERVENTIONS:
Procedure: Laser therapy — Erbium YAG laser

SUMMARY:
Patients seen with stress urinary incontinence (SUI) that have failed conservative treatments will be offered to participate in a sham controlled RCT of outpatient therapy with the Fotona Smooth Erbium Yag laser. Patients will be randomised to either outpatient laser treatments or sham treatments. Patients will be blinded to which arm they have been randomised. Patients will be asked to complete appropriate relevant symptom and quality of life questionnaires prior to treatment and then at 6 and 12 months following the final treatment. At 6 months Sham patients will be un-blinded and offered the laser therapy if they wish.

DETAILED DESCRIPTION:
All patients with urodynamically proven SUI, who have failed/declined conservative therapies and their history suggests mild to moderate SUI, will be informed about the study and consented if they wish.

They will be invited to attend a screening visit. At this visit, they will be asked to perform a standardised 1 hour pad test. Their medical history will be checked and they will undergo a clinical and vaginal examination, pregnancy test and dip stick urinalysis.If their 1 hour pad weight is >2g and <25g and they meet all other inclusion / exclusion criteria, they will be eligible for inclusion.

At the Baseline visit, the patient will have medical history confirmed, and be asked to complete a standing and supine (lying) cough test. They will be given the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) and Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) questionnaire. Patients will be randomised using a computer randomisation programme and blinded to their allocated arm: active treatment or sham treatment.

Patients will then undergo 3 outpatient treatment visits. The timing of visits will be 1 month apart. At each visit they will be asked if they have any further questions and if they are happy to continue to participate in the study. If happy to participate, they will have their urine tested for infection (dipstick urinalysis) and pregnancy test at each treatment appointment. If urinalysis is negative, they will receive an outpatient Incontilase laser treatment. At each of their 3 outpatient appointments, they will be asked about any deleterious effects since their last appointment and asked to complete an ICIQ-SF and Patient Global Impression of Improvement questionnaire (treatment 2 onwards). Patients will receive 3 treatments in total.

Patients will be invited to attend a follow up visits 6 & 12 months after the 3rd treatment and asked to complete ICIQ-SF, PISQ-12 and PGI-I symptom questionnaires and undergo a clinical examination. They will be asked to perform a cough test supine (lying) and standing and at 6 and 12 months also perform a 1 hour pad test as described earlier (see appendices). Patients randomised to the Sham arm will be un-blinded at 6 months and offered the treatment if they wish and followed up for six months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Female, 18 years of age or older
2. Clinical and UDS diagnosis of Stress Urinary Incontinence
3. SUI on 1-hour Pad weight test between 2g and 25g (SUI I: 2-10g, SUI II:11-25g)
4. No significant improvement in urinary incontinence from at least one previous conservative treatment, such as pelvic floor muscle training

Exclusion Criteria:

1. Pre-existing bladder pathology including prior radiation treatment
2. Pregnancy
3. BMI>35
4. Radical pelvic surgery or previous incontinence surgery
5. Urinary tract infection or other active infections of urinary tract or bladder
6. SUI on 1 hour pad weight test >25g (SUI III: >25g)
7. Any form of pelvic organ prolapse greater than stage 2, according to POP-Q
8. Diagnosis of urge incontinence
9. Diagnosis of collagen disorders eg.benign joint hypermobility / Elhers-Danlos / Marfans etc.
10. Incomplete bladder emptying
11. Vesicovaginal fistula
12. Faecal incontinence
13. Unwillingness or inability to complete follow-up schedule
14. Unwillingness or inability to give Informed Consent
15. Failure to comply with diary requirements during extended baseline period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of 1hr pad weight test | 6 months
  The change in standardised 1hr pad weight test from baseline to 6 months following treatment compared with the sham arm.

SECONDARY OUTCOMES:
Change in cough stress test from baseline to 6 months post treatment | 6 months
  change in cough stress test (positive or negative, ie urine leakage or no leakage)
Change in cough stress test from baseline to 12 months post treatment | 12 months
  change in cough stress test (positive or negative, ie urine leakage or no leakage)
change in 1-hour pad weight test from baseline to 12 months post treatment | 12 months
  change in 1-hour pad weight test (urine leakage over 1hr measured in g)
International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) from baseline to 6 months post treatment | 6 months
  Change in mean test scores range = 0 - 21; low score = mild symptoms, high score = significant impact on quality of life
International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) from baseline to 12 months post treatment | 12 months
  Change in mean test scores range = 0 - 21; low score = mild symptoms, high score = significant impact on quality of life
Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) from baseline to 6 months post treatment | 6 months
  Change in mean test scores range = 0 - 48; Higher value = increased sexual function, lower value = less sexual function
Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) from baseline to 12 months post treatment | 12 months
  Change in mean test scores range = 0 - 48; Higher value = increased sexual function, lower value = less sexual function
Patient's Global Impression of Improvement (PGII) at 6 months post treatment | 6 months
  Assessments of patients' outcome of treatment; range 1 - 7; range 1 (very much worse) to 7 (very much improved)
Patient's Global Impression of Improvement (PGII) at 12 months post treatment | 12 months
  Assessments of patients' outcome of treatment; range 1 - 7; range 1 (very much worse) to 7 (very much improved)
Pain visual analogue scale | 3 months
  Patient reported assessment of pain on 10cm visual analogue scale during treatment, range 0 - 10cm; 0= no pain, 10= severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Christian Phillips, Principal Investigator — Hampshire Hospitals NHS Foundation Trust
Locations (1):
- Basingstoke & North Hampshire Hospital, Basingstoke, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phillips C, Shah G, Gamper M, Kuszka A, Chandrakumaran K, Viereck V. Vaginal Erbium Laser for the Treatment of Mild-to-Moderate Stress Urinary Incontinence: A Multicentre Randomised Sham-Controlled Trial. BJOG. 2025 Nov 12. doi: 10.1111/1471-0528.70080. Online ahead of print. PMID 41221700
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601